CLINICAL TRIAL: NCT06845956
Title: Prevalence, Clinical Features, and Prognosis of Coronary Artery Embolism With Concomitant Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Ningbo University (Network)
Responsible Party: Principal Investigator, Jinsong Cheng，MD, Doctor of medicine, Chief physician, First Affiliated Hospital of Ningbo University
Other Study IDs: Project No. 213RS, 2024; Grant No 2022L001 (Other Grant/Funding Number: Ningbo Clinical Research Center for Cardiovascular Disease); 2021C03096 (Other Grant/Funding Number: Key research and development project of Zhejiang Province, China)
Record Dates: First submitted 2024-11-29; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Coronary Artery Embolism; Acute Myocardial Infarction Type 2
Keywords: coronary artery ebolism; acute myocardial infarction; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- coronary artery embolism with concomitant atrial fibrillation: myocardial infarction patients who were coronary artery embolism with concomitant atrial fibrillation
- Non-CE myocardial infarction with concomitant atrial fibrillation: myocardial infarction with concomitant atrial fibrillation(Non-coronary artery embolism )
- myocardial infarction without concomitant atrial fibrillation: myocardial infarction without concomitant atrial fibrillation without coronary artery embolism
  Interventions: Other: Is it coronary artery embolism

INTERVENTIONS:
Other: Is it coronary artery embolism — This observational study categorizes patients with acute myocardial infarction (AMI) into three distinct groups based on their clinical characteristics:
  1. Group 1: Patients with atrial fibrillation (AF) and coronary artery embolism (CAE).
  2. Group 2: Patients with AF but non-coronary artery embolism myocardial infarction (non-CAE MI).
  3. Group 3: Patients without AF and non-coronary artery embolism myocardial infarction (non-CAE MI without AF).
  A key innovation of this study compared to previous research is its expanded eligibility criteria for AMI patients. Earlier studies typically focused exclusively on ST-segment elevation myocardial infarction (STEMI). In contrast, this investigation encompasses a broader spectrum of acute myocardial infarction, including both STEMI and non-ST-segment elevation myocardial infarction (NSTEMI). This comprehensive approach enhances the generalizability and applicability of the findings by capturing a wider range of clinical scenarios.
  Groups: myocardial infarction without concomitant atrial fibrillation

SUMMARY:
The goal of this observational study is to learn about the Prevalence, Clinical Features, and Prognosis of Coronary Artery Embolism With Concomitant Atrial Fibrillation. The main question it aims to answer is:

What is the proportion of coronary artery embolism with concomitant atrial fibrillation among all myocardial infarctions and myocardial infarctions with concomitant atrial fibrillation? What are the clinical characteristics of coronary artery embolism with concomitant atrial fibrillation? What is the prognosis of coronary artery embolism with concomitant atrial fibrillation? All participants will receive routine diagnosis and treatment, and baseline demographic data, clinical examination laboratory results, and follow-up data will be collected for analysis.

DETAILED DESCRIPTION:
The study is designed as an observational study without involving experimental drugs or device interventions, only collecting data from routine medical practice.

Importance: Atrial fibrillation (AF) and acute myocardial infarction (AMI) share common risk factors and interact pathophysiologically. Coronary embolism (CE) is a critical mechanism of AMI in AF patients, yet its clinical features and prognosis remain understudied.

Objective: To investigate the incidence, clinical characteristics, and prognosis of CE in patients with AF.

Design, Setting, and Participants: A single-center retrospective case-control study was conducted at the Affiliated First Hospital of Ningbo University, China. Patients diagnosed with AMI who underwent coronary angiography (CAG) between January 1, 2014, and December 31, 2023, were included. CE was diagnosed using the Shibata criteria. Participants were categorized into three groups: AF-related CE, non-CE AF with AMI, and AMI without AF.

Main Outcomes and Measures: Baseline characteristics, clinical features, coronary involvement, treatment strategies, and outcomes (all-cause mortality, cardiac-death mortality, major adverse cardiovascular and cerebrovascular events [MACCE], recurrent embolism, and major bleeding) were compared.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Acute myocardial infarction
* Selective coronary angiography has been performed.

Exclusion Criteria:

* Clinical diagnosis of Iatrogenic coronary artery embolism
* Clinical diagnosis of Coronary artery dilation
* Clinical diagnosis of Coronary in-stent thrombosis and embolism
* Clinical diagnosis of Coronary slow flow syndrome
* Clinical diagnosis of Coronary artery dissection
* Clinical diagnosis of Coronary artery spasm
* Pathological examination showed that the embolus contained atherosclerotic plaque
* Endovascular imaging examinations, including intravascular ultrasound (IVUS) and optical coherence tomography (OCT), indicate the presence of plaque rupture, erosion, or ulceration in the culprit vessel.
* Clinical diagnosis of Previous myocardial infarction
* Previous coronary stent implantation or coronary artery bypass surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute myocardial infarction, with a history of atrial fibrillation or presenting with atrial fibrillation upon admission, who have undergone selective coronary angiography confirming typical thromboembolic events, with imaging studies identifying the thrombus origin from the left atrial appendage, with or without associated systemic embolism.
Sampling Method: Probability Sample
Enrollment: 5163 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
All-cause death, cardiogenic death | Up to 10 years
Major Adverse Cardiovascular and Cerebrovascular Events | Up to 10 years
Systemic thrombo-embolism | Up to 10 years
  Brain embolism, lower extremity arterial embolism, mesenteric arterial embolism, coronary artery embolism, splenic embolism, renal embolism.
Major hemorrhage | Up to 10 years
  BARC Grades 3-5 Bleeding

CONTACTS AND LOCATIONS:
Overall Officials: CUI H bin, Doctor, Study Director — Key research and development project of Zhejiang Province,Ningbo Clinical Research Center for Cardiovascular Disease
Locations (2):
- China (2):
  - The First affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tsao CW, Aday AW, Almarzooq ZI, Anderson CAM, Arora P, Avery CL, Baker-Smith CM, Beaton AZ, Boehme AK, Buxton AE, Commodore-Mensah Y, Elkind MSV, Evenson KR, Eze-Nliam C, Fugar S, Generoso G, Heard DG, Hiremath S, Ho JE, Kalani R, Kazi DS, Ko D, Levine DA, Liu J, Ma J, Magnani JW, Michos ED, Mussolino ME, Navaneethan SD, Parikh NI, Poudel R, Rezk-Hanna M, Roth GA, Shah NS, St-Onge MP, Thacker EL, Virani SS, Voeks JH, Wang NY, Wong ND, Wong SS, Yaffe K, Martin SS; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2023 Update: A Report From the American Heart Association. Circulation. 2023 Feb 21;147(8):e93-e621. doi: 10.1161/CIR.0000000000001123. Epub 2023 Jan 25. PMID 36695182
- [Background] Shibata T, Kawakami S, Noguchi T, Tanaka T, Asaumi Y, Kanaya T, Nagai T, Nakao K, Fujino M, Nagatsuka K, Ishibashi-Ueda H, Nishimura K, Miyamoto Y, Kusano K, Anzai T, Goto Y, Ogawa H, Yasuda S. Prevalence, Clinical Features, and Prognosis of Acute Myocardial Infarction Attributable to Coronary Artery Embolism. Circulation. 2015 Jul 28;132(4):241-50. doi: 10.1161/CIRCULATIONAHA.114.015134. Epub 2015 Jun 25. PMID 26216084
- [Background] Menke J, Luthje L, Kastrup A, Larsen J. Thromboembolism in atrial fibrillation. Am J Cardiol. 2010 Feb 15;105(4):502-10. doi: 10.1016/j.amjcard.2009.10.018. PMID 20152245
- [Background] Popovic B, Varlot J, Humbertjean L, Sellal JM, Pace N, Hammache N, Fay R, Eggenspieler F, Metzdorf PA, Camenzind E. Coronary Embolism Among Patients With ST-Segment-Elevation Myocardial Infarction and Atrial Fibrillation: An Underrecognized But Deadly Association. J Am Heart Assoc. 2024 May 21;13(10):e032199. doi: 10.1161/JAHA.123.032199. Epub 2024 May 14. PMID 38742522
- [Background] Jia H, Abtahian F, Aguirre AD, Lee S, Chia S, Lowe H, Kato K, Yonetsu T, Vergallo R, Hu S, Tian J, Lee H, Park SJ, Jang YS, Raffel OC, Mizuno K, Uemura S, Itoh T, Kakuta T, Choi SY, Dauerman HL, Prasad A, Toma C, McNulty I, Zhang S, Yu B, Fuster V, Narula J, Virmani R, Jang IK. In vivo diagnosis of plaque erosion and calcified nodule in patients with acute coronary syndrome by intravascular optical coherence tomography. J Am Coll Cardiol. 2013 Nov 5;62(19):1748-58. doi: 10.1016/j.jacc.2013.05.071. Epub 2013 Jun 27. PMID 23810884
- [Background] Frederiksen TC, Dahm CC, Preis SR, Lin H, Trinquart L, Benjamin EJ, Kornej J. The bidirectional association between atrial fibrillation and myocardial infarction. Nat Rev Cardiol. 2023 Sep;20(9):631-644. doi: 10.1038/s41569-023-00857-3. Epub 2023 Apr 17. PMID 37069297
- [Background] Obayashi Y, Shiomi H, Morimoto T, Tamaki Y, Inoko M, Yamamoto K, Takeji Y, Tada T, Nagao K, Yamaji K, Kaneda K, Suwa S, Tamura T, Sakamoto H, Inada T, Matsuda M, Sato Y, Furukawa Y, Ando K, Kadota K, Nakagawa Y, Kimura T; CREDO-Kyoto AMI Registry Wave-2 Investigators. Newly Diagnosed Atrial Fibrillation in Acute Myocardial Infarction. J Am Heart Assoc. 2021 Sep 21;10(18):e021417. doi: 10.1161/JAHA.121.021417. Epub 2021 Sep 17. PMID 34533047
- [Background] Lee JH, Kim SH, Lee W, Cho Y, Kang SH, Park JJ, Oh IY, Yoon CH, Suh JW, Cho YS, Youn TJ, Chae IH, Choi DJ. New-onset paroxysmal atrial fibrillation in acute myocardial infarction: increased risk of stroke. BMJ Open. 2020 Sep 23;10(9):e039600. doi: 10.1136/bmjopen-2020-039600. PMID 32967885
- [Background] Vaduganathan M, Mensah GA, Turco JV, Fuster V, Roth GA. The Global Burden of Cardiovascular Diseases and Risk: A Compass for Future Health. J Am Coll Cardiol. 2022 Dec 20;80(25):2361-2371. doi: 10.1016/j.jacc.2022.11.005. Epub 2022 Nov 9. No abstract available. PMID 36368511